CLINICAL TRIAL: NCT01557309
Title: Arthroscopic Repair of Traumatic Rotator Cuff Tears. A Prospective Trial
Brief Title: Clinical and Structural Outcome After Early Repair of the Traumatic Rotator Cuff Tear
Status: Completed | Type: Observational
Sponsor: Helsingborgs Hospital (Other)
Responsible Party: Principal Investigator, Knut Aagaard, MD, MD., Lund University
Other Study IDs: KAstudy2
Record Dates: First submitted 2012-01-27; First posted 2012-03-19 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Full Thickness Rotator Cuff Tear
Keywords: traumatic rotator cuff tear; arthroscopic rotator cuff repair; age; early rotator cuff repair

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peroperatively retained rotator cuff biopsy.

SUMMARY:
The optimal timing for surgical repair of traumatic rotator cuff tears is controversial. Today there are no prospective studies investigating the short to mid-term outcome after early arthroscopic repair of traumatic rotator cuff tears and the Swedish National Musculoskeletal Competence Centre requests more research to this subject. The investigators will follow 60 patients with acute rotator cuff tear undergoing early rotator cuff repair during the first year after surgery.

The investigators hypothesise that the outcome after rotator cuff repair is good.

DETAILED DESCRIPTION:
There exists controversy in the current literature regarding timing for surgical repair of traumatic rotator cuff tears. We have seen no prospective studies describing the progression of shoulder function improvement the first year after arthroscopic rotator cuff repair.

We hypothesize that early arthroscopic repair of traumatic rotator cuff tears yields successful functional and structural outcomes but there will be a progression of shoulder function improvement during the hole first postoperative year.

ELIGIBILITY:
Inclusion Criteria:

* trauma to the shoulder with sudden onset of symptoms
* asymptomatic shoulder before trauma
* mr positive for full thickness rotator cuff tear

Exclusion Criteria:

* fracture
* severe comorbidity
* more than 6 weeks after trauma
* glenohumeral degeneration signs or osteoarthritis on x-ray

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective trial analysing the results after early arthroscopic repair of the traumatic rotator cuff tear. Every consecutive patient between Nov 2010 and Oct 2013 who fulfill the inclusion criteria are asked to participate after oral and written information. With a population of 250.000 we approximate an enrollment of 60 participants.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-11; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Western Ontario Rotator Cuff Index (WORC) | Two years

SECONDARY OUTCOMES:
Constant Shoulder Score (CS) | One year
standardised measure of health status with EQ-5D | Two years
cuff integrity | One year
Complications | within one year

CONTACTS AND LOCATIONS:
Overall Officials: Karl Lunsjo, Ass Prof, Study Director — Helsingborgs Hospital
Locations (1):
- Department of Orthopaedic Surgery, Helsingborg Hospital, Helsingborg, Sweden

REFERENCES:
- [Background] Bassett RW, Cofield RH. Acute tears of the rotator cuff. The timing of surgical repair. Clin Orthop Relat Res. 1983 May;(175):18-24. PMID 6839586
- [Background] Lahteenmaki R, Lawrence S. Public biotech 2006 - the numbers. Nat Biotechnol. 2007 Jul;25(7):729-37. doi: 10.1038/nbt0707-729. No abstract available. PMID 17621294
- [Background] Bjornsson HC, Norlin R, Johansson K, Adolfsson LE. The influence of age, delay of repair, and tendon involvement in acute rotator cuff tears: structural and clinical outcomes after repair of 42 shoulders. Acta Orthop. 2011 Apr;82(2):187-92. doi: 10.3109/17453674.2011.566144. Epub 2011 Mar 24. PMID 21434791
- [Background] Petersen SA, Murphy TP. The timing of rotator cuff repair for the restoration of function. J Shoulder Elbow Surg. 2011 Jan;20(1):62-8. doi: 10.1016/j.jse.2010.04.045. Epub 2010 Aug 1. PMID 20675154
- [Background] Sorensen AK, Bak K, Krarup AL, Thune CH, Nygaard M, Jorgensen U, Sloth C, Torp-Pedersen S. Acute rotator cuff tear: do we miss the early diagnosis? A prospective study showing a high incidence of rotator cuff tears after shoulder trauma. J Shoulder Elbow Surg. 2007 Mar-Apr;16(2):174-80. doi: 10.1016/j.jse.2006.06.010. Epub 2006 Dec 13. PMID 17169582
- [Background] Nho SJ, Adler RS, Tomlinson DP, Allen AA, Cordasco FA, Warren RF, Altchek DW, MacGillivray JD. Arthroscopic rotator cuff repair: prospective evaluation with sequential ultrasonography. Am J Sports Med. 2009 Oct;37(10):1938-45. doi: 10.1177/0363546509335764. Epub 2009 Jun 16. PMID 19531660